CLINICAL TRIAL: NCT04575077
Title: The Role of Hepcidin as a Biomarker to Predict Successful Renal Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-0748
Record Dates: First submitted 2020-09-18; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High hepcidin concentrations indicate that iron is blocked from secretion from the reservoir. Hepcidin may be useful in prediction functional iron utilization in renal failure patients. Hepcidin is also associated with chronic renal failure and residual renal function in dialysis patients. Recent studies have shown that hepcidin is a potential marker of impaired renal function in a rat model of chronic nephropathy.

The purpose of this study was to investigate the relationship between preoperative hepcidin levels and the incidence of success rate of kidney transplantation in patients with end-stage renal failure undergoing kidney transplantation surgery. The study is a prospective single-group observational study that analyzes hepcidin as a biomarker.

DETAILED DESCRIPTION:
POD-1 : Researchers will meet patients scheduled for surgery and explain the study. (enroll) the operation date : The patient will sign the consent form. Researchers will collect the blood sample from the patient for testing hepcidin during the operation and record laboratory data performed before surgery POD 1: laboratory test discharge date : laboratory test 6 months after surgery ; Researchers will determine the graft failure of the patient.

* laboratory test ; reticulocyte count, Hb, plasma hepcidin, iron profiles (serum iron, serum ferritin, total iron-binding capacity, transferrin, transferrin saturation), coagulation profiles (PT, PTT), routine urinary analysis, and chemical profiles (aspartate aminotransferase (AST)/alanine aminotransaminase (ALT), serum creatinine, electrolytes, C-reactive protein (CRP), estimated glomerular filtration rate (GFR)), ESR, cystatin C, NGAL, pro BNP, troponin T and urinary analysis

ELIGIBILITY:
Inclusion Criteria:

1. The patients who plan to undergo kidney transplantation
2. ASA III-IV
3. adult over 19 years old

Exclusion Criteria:

1. emergent case
2. heart disease
3. arrhythmia
4. BMI >30kg/m2
5. allergy to some drugs
6. if other co-operation is planned
7. foreigner
8. Illiteracy

Ages: 19 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage kidney disease who are expected to undergo kidney transplantation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | 6 months
  AKIN Criteria have only three stages of AKI (Stages I-III) which generally correspond to RIFLE stages R, I, and F. The AKIN group claims an advantage over the RIFLE criteria in that it has a lower threshold for defining an individual as Stage I AKI (only 0.3 mg/dL increase OR a 1.5X increase over baseline is required to meet this definition in AKIN; in RIFLE one requires a 1.5X increase over baseline. Both definitions can also be met by urine output criteria as well.)

SECONDARY OUTCOMES:
numbers of participants with abnormal laboratory values | 1) 1 month before the surgery, 2) Postoperative day(POD) 1, 3) 2 weeks after the surgery
  Laboratory test(reticulocyte count, Hb, plasma hepcidin, iron profiles (serum iron, serum ferritin, total iron-binding capacity, transferrin, transferrin saturation), coagulation profiles (PT, PTT), and chemical profiles (aspartate aminotransferase (AST)/alanine aminotransaminase (ALT), serum creatinine, electrolytes, C-reactive protein (CRP), estimated glomerular filtration rate (GFR)), ESR, cystatin C, NGAL, pro BNP, troponin T), routine urinary analysis
the number of participants with wound infection | 6 months after surgery
major adverse cardiac event | 6 months after surgery
the number of participants who hospitalize again | 6 months after surgery
mortality | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Nyeo Koo, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No